CLINICAL TRIAL: NCT06801028
Title: Efficacy of Injection Sekucinumab in Erythrodermic Psoriasis
Status: Not yet recruiting | Type: Observational
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Maria Iqbal, Primary investigator, MBBS, FCPS Trainee, Jinnah Postgraduate Medical Centre
Other Study IDs: NO.F.2-81/2024-GENL/137/JPMC
Record Dates: First submitted 2025-01-16; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Erythrodermic Psoriasis
Keywords: Erythrodermic Psoriasis; Efficacy; Sekucinumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Erythrodermic Psoriasis: Erythrodermic Psoriasis will be treated by injection Sekucinumab
  Interventions: Biological: injection Sekucinumab

INTERVENTIONS:
Biological: injection Sekucinumab — All patients with erythrodermic psoriasis (EP), who will receive subcutaneous injection of secukinumab at a dose of 300 mg once a week from week 0 to 4 followed by every 4 week. At weeks 0, 4, 8, 12, 16 and 20 the psoriasis area and severity index (PASI) will be recorded and adverse drug reactions, patient's satisfaction and recurrence will be observed.

SUMMARY:
Erythroderma is a rare and severe dermatological manifestation of a variety of diseases. The most common form of erythroderma is erythrodermic psoriasis (EP), which accounts for 1-2.25% of all psoriatic patients, with a male predominance as demonstrated by a male to female ratio of 3:1. EP clinically manifests with diffuse erythema involving also skin folds with or without exfoliate dermatitis. Secukinumab is a FDA approved biological targeting interleukin-17A (IL17A) cytokine used in the treatment of moderate-to-severe psoriasis. Many clinical trials have been undertaken to establish its efficacy and safety in psoriasis. Numerous studies have highlighted the efficacy and safety of secukinumab. Secukinumab yields rapid and sustained improvements of signs and symptoms in patients EP. Secukinumab also had the lowest treatment cost compared with other biologic treatments for moderate to severe psoriasis. Secukinumab is a monoclonal antibody targeting IL-17, a key player in psoriasis pathogenesis, making it highly effective for psoriasis management. Erythrodermic psoriasis (EP) is a rare, severe form of the disease, affecting over 90% of the body, with significant health risks like electrolyte imbalance and infection. Treatment options for EP are not standardized due to its rarity, and conventional therapies such as acitretin, ciclosporin, and methotrexate have limited efficacy and tolerance issues. While biologics are well-studied for plaque psoriasis, data on EP is scarce. This study aims to evaluate secukinumab's efficacy in EP and explore factors influencing treatment outcomes.

DETAILED DESCRIPTION:
This observational descriptive longitudinal study will be conducted at OPD patients in the Department of Dermatology, Jinnah Postgraduate Medical Center. after taking ethical approval from institutional ethical review board. Informed consent will be obtained from all the patients. Erythrodermic Psoriasis patients aged 18 years and older, who received the complete treatment course of secukinumab will be included. Before secukinumab treatment, all infections including hepatitis B and C virus infection and tuberculosis (Tb) status are evaluated by history, physical examination, complete blood count, C reactive protein, transaminases, complete urinalysis, chest X-Ray studies, Purified Protein Derivative (PPD) test and/or QuantiFERON-TB tests and hepatitis B, C viruses markers, etc.

All patients with erythrodermic psoriasis (EP), who will receive subcutaneous injection of secukinumab at a dose of 300 mg once a week from week 0 to 4 followed by every 4 week. At weeks 0, 4, 8, 12, 16 and 20 the psoriasis area and severity index (PASI) will be recorded and adverse drug reactions, patient's satisfaction and recurrence will be observed.

Demographics and clinical features will be recorded, including: age; gender; previous Psoriasis Area Severity Index (PASI) score before erythroderma, if any; previous anti-psoriatic therapy; biologic therapy exposure; secukinumab response; side effects; drug use history; PASI and patients satisfaction at weeks 4, 8, 12, 16, and 20. Efficacy assessment will be performed by measuring change in PASI score from baseline. PASI-75 will be considered as efficacy of treatment. It will be assessed after treatment induction (Week 4) at 4, 8, 12, 16 and 20 week. Adverse effects, recurrence and reasons for discontinuation secukinumab will be recorded.

ELIGIBILITY:
Inclusion criteria:

* Patients of age 18-65 years age.
* Either sex.
* Patients presenting with the clinical manifestations of Erythrodermic Psoriasis such as redness, inflammation, skin rash, erythema, scaling, and itch on more than 90% of body surface area.

Exclusion criteria:

* Patients of pediatric age.
* Erythroderma caused by a condition other than psoriasis.
* Patient treated with biologics for a different condition other than EP.
* Diabetic, immunocompromised patients.
* Women with pregnancy or lactating mothers.
* Patients allergic to the drugs in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: EP Patients presenting with the histological and/or clinical manifestations (Erythrodermic Psoriasis such as redness, inflammation, skin rash, erythema, scaling, and itch) on more than 90% of body surface area.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy (Psoriasis Area Severity Index (PASI) Score) | 20th week
  The Psoriasis Area Severity Index (PASI) is an index used to express the severity of psoriasis.
  It combines the severity (erythema, induration and desquamation) and percentage of affected area. The Psoriasis Area Severity Index (PASI) Calculator (1.7.3) (https://pasi.corti.li/ ) or manual working sheet https://www.huidziekten.nl/pdf/PASI-Psoriasis-Area-and-Severity-Index.pdf.) will be utilized to calculate the PASI score at each time interval.
  Efficacy assessment will be performed by measuring change in PASI score from baseline. PASI-75 (75% or greater improvement/ 75% or more reduction in PASI score) will be considered as efficacy of treatment. It will be assessed after treatment induction (Week 4) at 4, 8, 12, 16 and 20 week.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Iqbal, MBBS, FCPS Trainee, Principal Investigator — JPMC
Locations (1):
- Department of Dermatology Jinnah Postgraduate Medical Center (JPMC), Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No